CLINICAL TRIAL: NCT06203444
Title: An Open-label Study to Evaluate the Pharmacokinetics of Oral Tenapanor in Breast Milk of Lactating Females
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ardelyx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TEN-01-109
Record Dates: First submitted 2023-12-17; First posted 2024-01-12 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Lactation
MeSH Terms: conditions — Breast Feeding | interventions — tenapanor

STUDY DESIGN:
Intervention Model Description: An open-label study to investigate the PK of tenapanor and AZ13792925 in breast milk of lactating female subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Eligible subjects will be enrolled to receive the study drug
  Interventions: Drug: Tenapanor

INTERVENTIONS:
Drug: Tenapanor — The study drug will be administered in dose of 50 mg bid
  Other Names: IBSRELA

SUMMARY:
This is an open label study to investigate PK of tenapanor and AZ13792925 in breast milk of lactating female subjects.

DETAILED DESCRIPTION:
This will be an open-label study to investigate the PK of tenapanor and AZ13792925 in breast milk of lactating female subjects. Potential subjects will be screened to assess their eligibility to enter the study within 15 days prior to the first dose administration. Subjects will receive tenapanor from Days 1 to 4 and will be monitored for 24 hours after the last dose of tenapanor. On Day 4, breast milk to evaluate concentrations of tenapanor and AZ13792925 will be collected pre-dose (Hour 0), 1, 2, 4, 6, 8, and 24 hours post-dose. Subjects will return for a Follow-up visit, 5 to 7 days (Day 10±1) after the last dose. All breast milk not used for PK analyses will be discarded (not fed to infant) starting on Day 1 after the first dose of tenapanor is administered until Day 7 (72 hours after last dose of tenapanor).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must satisfy all of the following criteria at the Screening visit unless otherwise stated:

  1. Females greater than or equal to 18 years of age.
  2. Body mass index between 18.0 and 35.0 kg/m2, inclusive.
  3. In good health with no clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs measurements, and clinical laboratory as determined by the Investigator.
  4. Females must be non-pregnant.
  5. Has been breastfeeding or actively pumping for at least 4 weeks.
  6. Willing to continue regular pumping in order to maintain milk supply for the duration of the study.
  7. Will not feed infant breast milk while taking tenapanor and for 72 hours post the last dose of tenapanor.
  8. Weaning must not be underway, to ensure an adequate milk supply.
  9. Able to comprehend and willing to sign an ICF and to abide by the study restrictions

Exclusion Criteria:

Subjects will be excluded from the study if they satisfy any of the following criteria at the Screening visit unless otherwise stated:

1. Significant medical or psychiatric disorder, as determined by the Investigator that would interfere with participation.
2. Use or intend to use any prescription or non-prescription medications 4 days before first dose of tenapanor until Day 6 of the study, unless deemed acceptable by the Investigator and/or Sponsor.
3. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed).
4. Has mastitis or other condition that would prevent the collection of milk from one or both breasts.
5. Loose stools (Type 6 or 7 on the Bristol Stool Form Scale) ≥2 days in the past 7 days
6. Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 30 days prior to dosing or 5 half-lives prior to dosing.
7. Subjects who, in the opinion of the Investigator (or designee), should not participate in this study

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Lactating Females
Enrollment: 7 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Concentration of tenapanor and its major metabolite in breast milk | 26 Days
  The primary objective of the study is to determine the maximum observed milk concentration (Cmax) of tenapanor and its primary metabolite AZ13792925 in the breast milk of lactating female subjects.

SECONDARY OUTCOMES:
The safety of tenapanor in lactating females | 26 Days
  The secondary objective of the study is to assess the the incidence and severity of treatment-emergent adverse events of tenapanor when administered to lactating female subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Edelstein, PhD, Study Director — Ardelyx
Locations (2):
- United States (2):
  - DDSI, Oklahoma City, Oklahoma
  - Fortrea Clinical Research Unit, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No